CLINICAL TRIAL: NCT03162588
Title: Feasibility Study of Multiple Burrhole Therapy Combined With Intravenous Erythropoietin Pretreatment for Unstable Moyamoya
Brief Title: Multiple Burrhole Therapy With Erythropoietin for Unstable Moyamoya
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Man Hong, Associate Proffessor of Neurology, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-T12-11-065
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Ischemic Attack; Ischemic Stroke; Moyamoya Disease; Burr Hole; Angiogenesis
MeSH Terms: conditions — Ischemic Stroke; Moyamoya Disease | interventions — Erythropoietin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multiple burrhole therapy and erythropoietin (Experimental): pretreatment with IV erythropoietin for 3 days, 120000IU#3 then multiple burrhole procedure on the hemisphere effected is performed
  Interventions: Drug: erythropoietin

INTERVENTIONS:
Drug: erythropoietin — Epokine®, CJ healthcare, South Korea is used preprocedurally to promote revascularization. Total 120,000 units of EPO is injected for three consecutive days, 40,000 units mixed in IV saline 100 ml over 1 hour. The multiple burrhole procedure is performed in area of hemodynamic insufficiency by D-SPECT. It is performed under local anesthesia.
  Other Names: multiple burrhole procedure

SUMMARY:
In this study, the investigators aim to evaluate the indirect revascularization outcomes of a new combination therapy of multiple burrhole procedure with promotion of arteriogenesis by intravenous (IV) erythropoietin (EPO) pretreatment on Moyamoya patients with acute neurological presentation, and outline the clinical and vascular factors associated with revascularization through the burrholes.

DETAILED DESCRIPTION:
This is a investigator led, single-center, single arm, interventional trial in prospective Moyamoya disease (MMD) and Moyamoya syndrome (MMS) registry. MMD or MMS patients with acute neurological presentation such as ischemic stroke or transient ischemic attack are eligible.

After inclusion, initial evaluation including transfemoral angiography is performed. A 3 day pre-procedure IV erythropoietin (120000 international units[IU] #3) is given for promotion of arteriogenesis, than multiple burrhole procedure is performed. Arteriogenesis is evaluated by 6 month transfemoral angiography.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years
* Acute neurological presentation with recurrent transient ischemic attacks (TIA) or cerebral infarction within 30 days of symptom onset
* Angiographic findings compatible with the diagnostic criteria for MMD or MMS (unilateral findings, bilateral distal internal carotid artery involvement without Moyamoya vessels, or presence of other causative factors)
* Significant decrease in basal perfusion and reservoir capacity on brain perfusion CT or Brain single photon emission computed tomography with acetazolamide (Diamox®) challenge (D-SPECT)

Exclusion Criteria:

* Definite presence of transdural collateral flow on cerebral angiography.
* Sufficient perfusion status via Willisian, leptomeningeal, or other collateral systems, as evaluated by multimodal imaging methods.
* > 30 days after symptom onset

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Functional status of the participants after 6 months of procedure assessed by modified Rankin Scale. | 6 month post-procedure
  The functional status of participants will be assessed based on modified Rankin Scale for evaluation of feasibility of procedure.
transdural arteriogenesis | 6 month post-procedural cerebral angiography
  the extent of collateral flow that has developed from external carotid artery to internal carotid artery through the burrholes

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Any complications occuring within <14 days of burrhole procedure + erythropoietin is classified as periprocedural complications. Any complications occuring or detected after 14 days of procedure up to 6 months will be classified as post-procedural.
  periprocedural and post-procedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Ji Man Hong, Principal Investigator — assistant professor of neurology
Locations (1):
- Ajou University Medical Center, Suwon, Gyunggido, South Korea

REFERENCES:
- [Derived] Hong JM, Lee SJ, Lee JS, Choi MH, Lee SE, Choi JW, Lim YC. Feasibility of Multiple Burr Hole With Erythropoietin in Acute Moyamoya Patients. Stroke. 2018 May;49(5):1290-1295. doi: 10.1161/STROKEAHA.117.020566. Epub 2018 Apr 6. PMID 29626135